CLINICAL TRIAL: NCT06087848
Title: A Longitudinal Open-Label Multi-center Single-Arm Phase I/IIa Study to Evaluate the Safety and Preventive Effect on Cardiovascular Events of Human Allogenic Bone-Marrow-Derived Mesenchymal Stromal Cell Product, StromaForte, in Study Participants.
Brief Title: A Study to Evaluate Mesenchymal Stem Cell Product StromaForte's Effect on Cardiovascular Events
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellcolabs Clinical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-001-BHS
Record Dates: First submitted 2023-10-04; First posted 2023-10-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC Intervention Group (Experimental): Participants will receive 100 x 106 allogeneic bone marrow (BM)-derived Mesenchymal Stromal Cells in one intravenous infusion.
  Additional systemic treatments can be repeated after a minimum of 3 months and data will be collected to investigate the potential preventive benefits it provides for the above indications. Additional doses are optional for all study participants enrolled in the study and will be managed in a separate consenting process. Study participants opting for an extra dose must at the time of the extra dose meet the same inclusion and exclusion criteria as participants being included for the first dose
  Interventions: Biological: Human Allogeneic Bone-Marrow-Derived Mesenchymal Stromal Cell Product (StromaForte)

INTERVENTIONS:
Biological: Human Allogeneic Bone-Marrow-Derived Mesenchymal Stromal Cell Product (StromaForte) — 100 x 106 allogeneic bone marrow (BM)-derived Mesenchymal Stromal Cell (MSC) formulated in sodium chloride supplemented with human serum albumin to be given via slow intravenous infusion in approximately 30 min

SUMMARY:
The goal of this phase I/II clinical trial is to evaluate the safety and preventive effect of intravenous infusion of human allogeneic bone-marrow-derived mesenchymal stromal cell product StromaForte in study participants. The main questions it aims to answer are:

To assess the safety and tolerability after 28 days of injection by reporting the number of adverse events assessed by Common Terminology Criteria For Adverse Events (CTCAE) To evaluate the effects of Mesenchymal stem cells on Prevention of Cardiovascular Events by following the reported incidence of cardiovascular events amongst study participants up to five year post-injection Participants will receive 100 x 106 allogeneic bone marrow (BM)-derived Mesenchymal Stromal Cell (MSC) formulated in sodium chloride supplemented with human serum albumin to be given via slow intravenous infusion 100 million cells in approximately 30 min

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a group of disorders of the heart and blood vessels including, among other coronary heart, cerebrovascular, and peripheral arterial diseases that are difficult to reverse once clinically verified. According to the WHO, CVDs are the leading cause of death globally, taking an estimated 17.9 million lives each year. More than four out of five CVD deaths are due to heart attacks and strokes, and one third of these deaths occur prematurely in people under 70 years of age (1). The onset of CVD may seem binary for the individual patient, one day one is healthy and the next one has suffered an event such as a myocardial infarction or a stroke. Thereby a vast majority of the treatments are interventions when a cardiovascular event happens, and consequently preventative efforts are mostly secondary prevention oriented, and therapies are often reduced to a monitoring of symptoms.

However, while some people are genetically predisposed to develop CVDs, everyone is at risk. CVDs is a group of aging- related chronic diseases, similarly to diabetes and arthritis, with an earlier onset than an eventual cardiovascular event. The vascular pathophysiology leading up to the first CVD event has often been gradually developing asymptomatically over years, driven by among other things tissue inflammation, endothelial dysfunction, and increased blood pressure, before the individual becomes aware of it. It is widely shown that ageing related diseases, like CVDs, are a huge challenge for societies around the globe, and that these groups consume up to 70-80 % of healthcare resources. Thus, healthy longevity is not only of interest for the individual but to society as well. If we are to reach the UN Sustainable Development Goal (SGD) #3 - Good Health and Wellbeing, prevention of diseases at an earlier stage is thought to play a key role.

The concept of preventive medicine is in its prime but there is a need for more research and scientific evidence around how to foster healthy longevity by retarding or preventing, among other things, the chronic inflammation that often drives the development of ageing related diseases. Acknowledging the gradual development of CVD, not only secondary prevention but also primary preventative treatment is an interesting strategy to examine further. Stem cells hold promise for mitigating the risk factors and reducing the incidence of these major health conditions. Due to their anti-inflammatory, regenerative, and immunomodulatory effects MSCs are an especially interesting candidate of preventive treatments, i.e., even for individuals without clinical symptoms, since ageing related diseases and vascular degeneration are partly driven by inflammation accelerated or slowed down by individual lifestyle, comorbidities, inherited genetics, age, and many other factors.

The Mesoblast DREAM-HF study published in 2023, indicated that there may be a potential secondary preventative effect of MSC on CVD. Mesenchymal Precursor Cell (MPC) therapy with local injection in the heart muscle did not meet its primary and secondary endpoints but resulted in significant reduced risk for time-to-first Major Adverse Cardiac Event (MACE) defined as cardiovascular death, Myocardial Infarction (MI) or stroke over a mean follow-up of 30 months with the most benefit seen in patients with evidence of systemic inflammation. The study also demonstrated a strengthened heart function, which was measured by the left ventricular ejection fraction (LVEF) for patients receiving the treatment compared to the control group.

To investigate the preventive, mitigating, and/or retarding effects of MSCs for the gradual disease development and/or degeneration across multiple cohorts of different risks this study is designed to follow a large and diverse study participant population over a long period of time (five years). All enrolled study participants will be risk stratified and categorized into different cohorts based on the well-established cardiovascular risk assessment tool Atherosclerotic Cardiovascular Disease (ASCVD) Risk calculator developed by American College of Cardiology and complementary questionnaires. All enrolled study participants will receive an initial dose of 100 x 106 MSCs that can be repeated at a minimum interval of 3 months. The endpoints collected from enrolled study participants will be compared to baseline as well as with the expected rates/outcomes from risk matched cohorts/patients in relevant open label registries (Real World Data - RWD) across the globe.

The study will assess changes in study participants' risk and life/lifestyle (based on the gold standards) from baseline throughout the study to account for external factors that might impact the disease's development. The study will also identify subgroups of study participants based on the number of doses received and the treatment frequency to assess the potential cumulative effects of the MSCs to provide new insights around host and dose response. To have a rich dataset and a more accurate comparison to cohorts in other registries, the ambition is to include data from follow-up visits and, by written consent from the study participants, study participants own general medical records, health scans and additional blood works. Ultimately, this study seeks to investigate the safety and efficacy of MSC therapy for preventing cardiovascular diseases by comparing individuals of the same risk-level that have received a MSC treatment against matched controls from RWD

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and comply with all procedures required by the protocol.
2. Aged ≥ 25 to 85 years at the time of signing the informed consent form.
3. Subjects with pre-morbid or stable morbid medical conditions, not requiring significant changes to their current medical therapy for > 6 months prior to enrolling in this study, are eligible

Exclusion Criteria:

1. Unwilling or unable to perform any of the assessments required by the protocol.
2. Have end stage liver or renal disease.
3. Have a clinical history of malignancy within 2.5 years (i.e., study participants with prior malignancy must be cancer free for 2.5 years) except curatively treated basal cell carcinoma, melanoma in situ, or cervical carcinoma.
4. Have any condition that limits lifespan to < 1 year according to the Principal Investigator's discretion.
5. Hepatitis B virus positive
6. Viraemic Hepatitis C virus, HIV-1/2 or syphilis positive
7. Have unstable angina pectoris, uncontrolled or severe peripheral artery disease within the previous 2 months.
8. Have congestive heart failure defined by New York Heart Association (NYHA) Class IV, or an ejection fraction of <25%.
9. Uncontrolled hypertension (resting systolic blood pressure >220 mm Hg or diastolic blood pressure of > 150 mm Hg at screening)
10. Have coronary artery bypass surgery, angioplasty, peripheral vascular disease revascularization, or a myocardial infarction within the previous month.
11. Have acute exacerbation of chronic obstructive lung disease stage III or IV (Gold classification), Have cognitive or language barriers that prohibit obtaining informed consent or any study elements.
12. Severe acute infection at time of screening and treatment with study drug
13. Pregnant or Breastfeeding
14. Currently participating (or participated within the previous 30 days of consent) in an investigational therapeutic or device trial.
15. Have a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the study participant's participation for the full duration of the study.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2029-10-06 (Estimated); Study Completion 2029-10-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the number of adverse events or severe adverse event assessed by Common Terminology Criteria For Adverse Events (CTCAE) of intravenous infusion of human allogeneic BM-derived MSCs product StromaForte for all study participants. | 28 day post-infusion
  To assess the safety of injection by reporting the number of adverse events or severe adverse event assessed by Common Terminology Criteria For Adverse Events (CTCAE) which is the Incidence of any treatment-emergent serious adverse events (TE-SAEs), defined as the composite of death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities determined per the Investigator's judgment.

SECONDARY OUTCOMES:
To evaluate the effects of MSCs on Prevention of Cardiovascular Events | From baseline to 5 years
  The secondary endpoint of this study is to evaluate the reported incidence of cardiovascular events among the study participants. Cardiovascular events include but are not limited to myocardial infarction (heart attack), stroke, coronary artery disease, heart failure, and peripheral arterial disease. By monitoring and documenting the occurrence of these events, the study aims to assess the impact of the intervention (e.g., treatment with mesenchymal stem cells) on reducing the overall burden of cardiovascular events in the study population.

OTHER OUTCOMES:
Incidence of Diabetes | From baseline to 5 years
  The exploratory endpoint of this study is to evaluate the reported incidence of diabetes among the study participants. By monitoring and documenting the occurrence of new cases of diabetes during the study period, the objective is to assess the potential influence of the intervention on the development or progression of diabetes in the study population.
Incidence of Arthritis | From baseline to 5 years
  The exploratory endpoint of this study is to evaluate the reported incidence of arthritis among the study participants. By monitoring and documenting the occurrence of new cases of arthritis during the study period, the objective is to assess the potential influence of the intervention on the development or progression of arthritis in the study population.
Changes in Blood Glucose levels | From baseline to 5 years
  Changes from baseline in Blood Glucose levels to 5 years
Changes in serum glucose levels | From baseline to 5 years
  Changes from baseline in serum glucose levels to 5 years
Changes in blood pressure levels both systolic and diastolic | From baseline to 5 years
  Changes from baseline in blood pressure both systolic and diastolic levels to 5 years
Changes in total cholesterol levels | From baseline to 5 years
  Changes from baseline in total cholesterol levels to 5 years
Changes in LDL cholesterol levels | From baseline to 5 years
  Changes from baseline in LDL cholesterol levels to 5 years
Changes in HDL cholesterol levels | From baseline to 5 years
  Changes from baseline in HDL cholesterol levels to 5 years
Changes in triglycerides levels | From baseline to 5 years
  Changes from baseline in triglycerides levels to 5 years
Changes in TNF-a | From baseline to 5 years
  Changes in TNF-a levels from baseline to 5 years
Changes in IL-6 | From baseline to 5 years
  Changes in IL-6 from baseline to 5 years
Changes in telomere length with qPCR methods | From baseline to 5 years
  Changes in telomere length with qPCR methods to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Live Well, Nassau, The Bahamas, The Bahamas

IPD SHARING:
Plan to Share IPD: Undecided